CLINICAL TRIAL: NCT06757413
Title: Virtual Reality Programme Incorporating Psychology and Physiotherapy for Chronic Low Back Pain: a Randomised Controlled Pilot Trial
Brief Title: Virtual Reality Programme Incorporating Psychology and Physiotherapy for Chronic Low Back Pain
Acronym: CLEVER-BODY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other); University of Valencia (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Chair Profesor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cardenal Herrera University 69; PID2020-115609RB-C22 (Other Grant/Funding Number: MINISTRY OF SCIENCE AND INNOVATION OF SPAIN)
Record Dates: First submitted 2024-12-20; First posted 2025-01-03 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: VIRTUAL REALITY; PHYSICAL ACTIVITY; Pain; Disability; Kinesophobia; Psychology
MeSH Terms: conditions — Motor Activity; Pain; Kinesiophobia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Virtual reality (Experimental): This study evaluates a 4-week multidisciplinary intervention for patients with chronic non-specific low back pain, combining physiotherapy and psychological approaches. Both components leverage virtual reality (VR) technology to address physical and psychological aspects of pain management, operating in parallel to maximize patient outcomes.
  Physiotherapy Component. The physiotherapy intervention consists of a therapeutic exercise program based on the principles of the "Back School," designed to improve strength, stability, mobility, and flexibility in the abdomino-lumbo-pelvic region and lower extremities. Over 8 sessions (2 per week), patients perform VR-guided exercises where visual-proprioceptive information is manipulated. The VR goggles alter the perceived degree of lumbar flexion and extension, creating a mismatch between actual and perceived movements to promote motor learning and reduce maladaptive movement patterns.
  Interventions: Other: Enhanced Virtual reality
- Control Group (treatment as usual) (Active Comparator): Participants will receive the usual treatment applied at the hospital.
  Interventions: Other: Active Comparator: Treatment as usual

INTERVENTIONS:
Other: Enhanced Virtual reality — This study evaluates a 4-week multidisciplinary intervention for patients with chronic non-specific low back pain, combining physiotherapy and psychological approaches. Both components leverage virtual reality (VR) technology to address physical and psychological aspects of pain management, operating in parallel to maximize patient outcomes. The physiotherapy intervention consists of a therapeutic exercise program based on the principles of the "Back School". Over 8 sessions (2 per week), patients perform VR-guided exercises where visual-proprioceptive information is manipulated.
  The psychological positive body image-based intervention consists of 4 sessions approaching 5 different clinical modules: Pain Psychoeducation, Body Awareness, Pain Acceptance, Body Appreciation and Functionality and Gratitude. 2 sessions (Body Awareness and Pain Acceptancce) will include virtual reality environments to enhance the clinical outcomes.
  Other Names: Virtual Reality Group; Experimental Group
  Arms: Enhanced Virtual reality
Other: Active Comparator: Treatment as usual — Participants will receive the usual treatment applied at the hospital
  Arms: Control Group (treatment as usual)

SUMMARY:
The main objective of this randomized controlled pilot trial is to investigate the efficacy of a 4-week multidisciplinary intervention for patients with chronic non-specific low back pain, combining a therapeutic exercise program in physiotherapy and a psychological intervention focused on positive body image in pain intensity, pain interference, emotional distress, kinesophobia and pain catastrophization. Both components are designed to operate in parallel over a 4-week period. The physiotherapy component consists of a therapeutic exercise program of 8 sessions, performed with virtual reality (VR) manipulating visual proprioceptive information during all lumbar movements in the different therapeutic exercises. The psychological positive body image-based intervention consists of 4 sessions approaching 5 different clinical modules: Pain Psychoeducation, Body Awareness, Pain Acceptance, Body Appreciation and Functionality and Gratitude. 2 sessions (Body Awareness and Pain Acceptancce) will include virtual reality environments to enhance the clinical outcomes.

DETAILED DESCRIPTION:
This study evaluates a 4-week multidisciplinary intervention for patients with chronic non-specific low back pain, combining physiotherapy and psychological approaches. Both components leverage virtual reality (VR) technology to address physical and psychological aspects of pain management, operating in parallel to maximize patient outcomes.

Physiotherapy Component The physiotherapy intervention consists of a therapeutic exercise program based on the principles of the "Back School," designed to improve strength, stability, mobility, and flexibility in the abdomino-lumbo-pelvic region and lower extremities. Over 8 sessions (2 per week), patients perform VR-guided exercises where visual-proprioceptive information is manipulated. The VR goggles alter the perceived degree of lumbar flexion and extension, creating a mismatch between actual and perceived movements to promote motor learning and reduce maladaptive movement patterns.

Exercises are performed in two sets, with intensity and repetitions individualized using the Borg 6-20 scale for Rating of Perceived Exertion (RPE). During the first two weeks, exercises are performed at an RPE of 14 without additional load, while in weeks three and four, intensity increases to an RPE of 15 with progressively added weights. This program aims to improve outcomes such as pain, disability, kinesiophobia, catastrophizing, quality of life, and physical fitness.

Psychological Component

The psychological intervention aims to enhance positive body image and emotional resilience while addressing pain interference and emotional distress. It consists of four weekly sessions, each lasting approximately one hour, structured as follows:

1. Session 1: Pain Psychoeducation. Participants learn about chronic pain, its influencing factors, and the role of body image, with an overview of the intervention modules.
2. Session 2: Body Awareness. A virtual reality body scan is introduced to increase awareness of body sensations and perceptions.
3. Session 3: Pain Acceptance. Participants explore strategies to accept pain and address variables contributing to chronic pain, such as paradoxical control and avoidance, using a VR environment.
4. Session 4: Body Appreciation and Gratitude. Exercises focus on fostering appreciation for body functionality and gratitude for its abilities.

Participants will first undergo eligibility screening and baseline assessments before starting the intervention. The study complies with the ethical principles outlined in the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with non-specific cLBP according to the COST B13 European guideline
* age older than 18
* an average pain score of 3 or higher on the 11-point Pain Numerical Rating Scale (PNRS-11; with 0 indicating no pain and 10 indicating the worst pain imaginable) in the 6 months prior.

Exclusion criteria:

* spinal tumour, infection, or fracture
* systemic disease
* fibromyalgia
* cauda equina syndrome
* previous spinal surgery
* musculoskeletal injuries in the lower extremities (e.g., sciatica or radiating lower extremity pain, numbness, or weakness symptoms).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Body Disability | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  Roland-Morris Questionnaire (RMQ) is a 24-item patient-reported outcome measure those inquiries about pain-related disability. Items are scored 0 if left blank or 1 if endorsed, for a total RMQ score ranging from 0 to 24.
Emotional Distress | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  The 4-item Brief Assessment of Distress about Pain (BADP) scale was developed to assess anxiety, fear, and depression related to pain, as well as an overall evaluation of distress about pain. Items are scored from 0 ("Not at all") to 4 ("Extreme"), for a total BADP score ranging from 0 to 16.
Pain Interference and Pain Intensity | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  The Brief Pain Inventory (BPI) scale was developed to assess the severity of pain and its impact on functioning. The scale consists of 9 items with qualitative and quantitative data on the following dimensions: "Worst pain in last 24 hours", "Least pain in last 24 hours", "Pain on average" and "Pain right now".
Health related Quality of life | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  The SF-12 Health Survey is a short, standardised questionnaire designed to assess people's health status and quality of life. It consists of 12 questions that evaluate 8 dimensions: physical functioning, limitations due to physical problems, bodily pain, general health, vitality, social functioning, limitations due to emotional problems, and mental health (anxiety and depression). Scores are reported on two scales: the Physical Component Summary (PCS) and the Mental Component Summary (MCS), each ranging from 0 to 100, with higher scores indicating better perceived physical and mental health.

SECONDARY OUTCOMES:
Fear of movement | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  The Tampa Scale for Kinesophobia (TSK-11SV) is an 11-item scale that measures kinesophobia with statements asking the subject to answer from 1 ("Strongly disagree"), to 4 ("Strongly agree").
Body Awareness | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a state-trait self-report questionnaire to measure multiple dimensions of interoception (awareness of bodily sensations). These dimensions have been chosen for their relationship to the intervention components and for their good psychometric quality. The scores range from 0 to 5, where higher scores indicate a higher level in that dimension.
Chronic Pain Acceptance | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  Chronic Pain Acceptance Questionnaire 8 (CPAQ-8). Numerical rating scale ranging from 0 "Never true" to 6 "Always true" where higher scores indicate a higher Chronic Pain Acceptance (Pain Willingness and Activity Engagement).
Body Appreciation | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  Body Appreciation Scale 2 (BAS-2) is a 10-item measure of one's acceptance, favorable opinions and respect of their own body with a numerical rating scale ranging from 1 "Never" to 5 "Always" where higher scores indicate a higher Appreciation of the body.
Appreciation of Body Functionality | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  Functionality Appreciation Scale (FAS). The scores range from 1 to 5, where higher scores indicate higher levels of appreciation of body functionality.
Pain Catastrophizing | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  The Pain Catastrophizing Scale (PCS) consists of 13 statements containing a number of thoughts and feelings typically present in the experience of pain. The items are divided into 3 categories: rumination, magnification and helplessness, with each item scored on a 5-point scale. The patient is asked to indicate the frequency with which these feelings or thoughts appear from 0 ("Not at all") to 4 ("All the time").
Depression | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  The Patient Health Questionnaire (PHQ-9). The scale is composed of 9 items to assess depressive symptoms and the patient is asked to indicate the frequency with which these feelings, thoughts or states appear from 0 ("Not at all) to 3 ("Nearly every day").
Anxiety | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  The Generalised Anxiety Disorder-7 (GAD-7) scale is composed of 7 items to assess the different dimensions of the Generalised Anxiety Disorder and the patient is asked to mark the frequency from 'Never' to 'almost every day' in the last two weeks.
Life satisfaction | Baseline (pre-intervention) and immediately post-intervention (at 4 weeks).
  The Satisfaction with Life Scale (SWLS) is a 5-item self-report tool measuring global life satisfaction-a cognitive component of subjective well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have to decide it between all the researchers

REFERENCES:
- [Background] Alleva JM, Diedrichs PC, Halliwell E, Peters ML, Dures E, Stuijfzand BG, Rumsey N. More than my RA: A randomized trial investigating body image improvement among women with rheumatoid arthritis using a functionality-focused intervention program. J Consult Clin Psychol. 2018 Aug;86(8):666-676. doi: 10.1037/ccp0000317. PMID 30035583
- [Background] Valenzuela-Moguillansky C, Reyes-Reyes A, Gaete MI. Exteroceptive and Interoceptive Body-Self Awareness in Fibromyalgia Patients. Front Hum Neurosci. 2017 Mar 13;11:117. doi: 10.3389/fnhum.2017.00117. eCollection 2017. PMID 28348526
- [Background] Bailey KA, Gammage KL, van Ingen C, Ditor DS. "It's all about acceptance": A qualitative study exploring a model of positive body image for people with spinal cord injury. Body Image. 2015 Sep;15:24-34. doi: 10.1016/j.bodyim.2015.04.010. Epub 2015 May 21. PMID 26002149
- [Background] Harvie DS, Broecker M, Smith RT, Meulders A, Madden VJ, Moseley GL. Bogus visual feedback alters onset of movement-evoked pain in people with neck pain. Psychol Sci. 2015 Apr;26(4):385-92. doi: 10.1177/0956797614563339. Epub 2015 Feb 17. PMID 25691362